CLINICAL TRIAL: NCT02140814
Title: Uncontrolled, Open Label, Pilot and Feasibility Study of Niacinamide in Polycystic Kidney Disease
Acronym: NIAC-PKD1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alan Yu, MB, BChir (Other)
Responsible Party: Sponsor-Investigator, Alan Yu, MB, BChir, Professor and Director, Kidney Institute, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000874
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Polycystic Kidney Disease
Keywords: PKD; niacinamide; Vitamin B3; Vitamin B
MeSH Terms: conditions — Polycystic Kidney Diseases | interventions — Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Niacinamide (Experimental): All subjects in this study will take niacinamide at a dose of 30 mg per kilogram of body weight by mouth daily, in two divided daily doses, for 12 months.
  Interventions: Dietary Supplement: Niacinamide

INTERVENTIONS:
Dietary Supplement: Niacinamide
  Other Names: Vitamin B3

SUMMARY:
The goal of this pilot study is to evaluate the feasibility of administering niacinamide to patients with autosomal dominant polycystic kidney disease, to develop methods to assess the biological efficacy of niacinamide, and to perform a preliminary exploration of its clinical effect on kidney cyst growth and kidney function.

DETAILED DESCRIPTION:
Niacinamide is a form of vitamin B3. Vitamin B3 is found in many foods including yeast, meat, fish, milk, eggs, green vegetables, beans, and cereal grains. Recent studies in mice have shown that niacinamide, at high doses, may slow kidney cyst growth from polycystic kidney disease (PKD).

By doing this study, the researchers will determine if a larger, long-term study to test whether niacinamide slows progression of PKD is justified.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of autosomal dominant polycystic kidney disease
* eGFR > 90ml/min/1.73m2 as determined from the serum creatinine by the CKD-EPI equation
* Ability to give informed consent in English

Exclusion Criteria:

* History of liver disease or abnormal liver function test
* Heavy alcohol intake
* Chronic diarrhea or malabsorption syndrome
* Thrombocytopenia
* Hypophosphatemia
* Pregnancy or lactation or plan to become pregnant during the study
* Treatment with anti-epileptic drugs
* Treatment with tolvaptan, current or within 2 months prior to screening
* Participation in another interventional trial currently or within 30 days prior to screening
* Partial or total nephrectomy or renal cyst reduction (including aspiration) done <1 year ago
* Cardiac pacemaker
* Presence of magnetic resonance-incompatible metallic clips (e.g. clipped cerebral aneurysm)
* Body weight >159 kg (350 lbs) or untreatable claustrophobia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Sirtuin deacetylase activity | Change from Baseline to 12 Months
  Assessed by the level of post-translational modifications of two intracellular markers (1. Acetylated and total p53 protein concentrations, 2. Phosphorylated and total retinoblastoma protein (Rb))

SECONDARY OUTCOMES:
Sirtuin deacetylase activity | Change from Baseline to 6 Months
  Assessed by the level of post-translational modifications of two intracellular markers (1. Acetylated and total p53 protein concentrations, 2. Phosphorylated and total retinoblastoma protein (Rb))
Estimated Glomerular Filtration Rate (eGFR) | 12 Months
  Measurements at each visit using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
Height-adjusted total kidney volumes (htTKV) | Change from Baseline to 12 Months
  Measurements will be taken from MRI images, and the annual percent change in htTKV will be compared to historical values reported in a separate study of a similar study population.
Biomarker levels | 12 Months
  Aliquots of the urine samples from visits to be tested for a panel of biomarkers related to cyst growth compared to baseline levels.
Subject pain | Change from Baseline to 12 Months
  Subject feelings collected via abbreviated pain questionnaire. Questionnaire will be used to calculate pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Yu, MB, BChir, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States